CLINICAL TRIAL: NCT01343550
Title: Creativity Group for Borderline Personality Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Robert Gregory, M.D., SUNY Upstate Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHS6019
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2011-02

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Borderline Personality; Borderline
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Creativity group for persons diagnosed with BPD (Experimental)
  Interventions: Other: creativity group

INTERVENTIONS:
Other: creativity group — This is a creativity group intervention. There will be 4 groups. Each group has one session per week. Each session is a duration of two hours.

SUMMARY:
The investigators hypothesize that a creativity skills group for Borderline Personality Disorder can reduce symptoms of BPD, depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* participant self-reports clinical diagnosis of Borderline Personality Disorder
* currently seeing an individual therapist on a regular basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Borderline Evaluation of Severity Over Time (BEST) | baseline, 5th week, post-intervention (week 8)

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | baseline, week 5, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Blake Bazel, M.S., Study Director — State University of New York - Upstate Medical University; Robbi Saletsky, Ph.D., Study Director — State University of New York - Upstate Medical University; Roger Greenberg, Ph.D., Study Director — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Background] Gunderson JG. Borderline personality disorder: ontogeny of a diagnosis. Am J Psychiatry. 2009 May;166(5):530-9. doi: 10.1176/appi.ajp.2009.08121825. PMID 19411380
- [Result] Jacob GA, Gabriel S, Roepke S, Stoffers JM, Lieb K, Lammers CH. Group therapy module to enhance self-esteem in patients with borderline personality disorder: a pilot study. Int J Group Psychother. 2010;60(3):373-87. doi: 10.1521/ijgp.2010.60.3.373. PMID 20590434